CLINICAL TRIAL: NCT02976350
Title: Multiple Hormone Deficiency Syndrome in Heart Failure With Preserved Ejection Fraction
Brief Title: Hormone Deficiency in Heart Failure With Preserved Ejection Fraction
Acronym: MHDS in HFpEF
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Antonio Cittadini, Clinical Professor, Federico II University
Other Study IDs: HormoneHFpEF001
Record Dates: First submitted 2016-05-14; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Heart Failure; Hormone Deficiencies
Keywords: Heart failure; Heart failure with preserved ejection fraction; GH deficiency; Testosterone deficiency; Low- T3 syndrome; Multiple Hormone Deficiencies
MeSH Terms: conditions — Heart Failure; Dwarfism, Pituitary; Euthyroid Sick Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — serum for determination of hormonal levels
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with HFpEF: Male patients with heart failure with preserved ejection fraction

SUMMARY:
The objective of this study is to describe the prevalence of Multiple Hormone Deficiencies in Heart Failure with preserved Ejection Fraction.

DETAILED DESCRIPTION:
Despite the effectiveness of the neurohormonal model to explain the progression of heart failure and the many insights that it provided for the development of new therapies, there is increasing clinical evidence that suggests that our current models fail to completely explain the disease progression. Thus, neurohormonal models may be necessary but not sufficient to explain all aspects of disease progression in the failing heart. There is evidence suggesting that in heart failure there is a metabolic imbalance characterized by the predominance of the catabolic status over the anabolic drive.

Consistent data coming from several independent groups have documented the reduced activity of most anabolic axes in HF with reduced ejection fraction. To date, no study has addressed the prevalence the presence and the prevalence of the Multiple Hormone Deficiencies in Heart Failure with preserved Ejection Fraction.

ELIGIBILITY:
Inclusion Criteria:

* Male patients of affected by CHF, secondary to ischemic or idiopathic dilated cardiomyopathy
* left ventricle ejection fraction > 50% or more

Exclusion Criteria:

* severe liver disease
* serum creatinine levels >2.5 mg/dl
* history of active cancer with life expectancy below 1 year acute coronary syndrome in the previous 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with stable chronic heart failure with preserved ejection fraction
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of Hormone deficiency | 1 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cittadini, Professor, Study Chair — Federico II University
Locations (1):
- Antonio Cittadini, Napoli, Italy

IPD SHARING:
Plan to Share IPD: Yes